CLINICAL TRIAL: NCT02893488
Title: A Phase I, Single Dose, Five-period Crossover Relative Bioavailability Study of a Fixed-dose Combination Dolutegravir/Abacavir/Lamivudine Dispersible Tablet as Compared to a Co-dose of TIVICAY and EPZICOM in Healthy Subjects
Brief Title: Relative Bioavailability Study of a Fixed-dose Combination Dolutegravir/Abacavir/Lamivudine Dispersible Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 200402
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: dolutegravir; abacavir; relative bioavailability; palatability; GSK2619619; palatability questionnaire; lamivudine; pediatric; calcium; dispersible tablet
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — abacavir, lamivudine drug combination; dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- SEQUENCE ABCDE (Experimental): Participants will receive treatment A in period 1, treatment B in period 2, treatment C in period 3, treatment D in period 4 and treatment E in period 5 (one treatment per period). Where A=EPZICOM (ABC 600 milligrams (mg)/3TC 300 mg) plus four TIVICAY (DTG 10 mg) tablets with zero mineral content (ZMC) water. B=Four TRIUMEQ (ABC 150mg/DTG 10 mg/3TC 75 mg) tablets dispersed in 40 milliliter (mL) stock solution 1 and consumed immediately. C=Four TRIUMEQ tablets dispersed in 40 mL stock solution 1, held for 30 minutes(mins), re-dispersed, and then consumed. D=Four TRIUMEQ tablets dispersed in 40 mL stock solution 2 and consumed immediately. E=Four TRIUMEQ tablets dispersed in 40 mL stock solution 2, held for 30 mins, re-dispersed, and then consumed.
  Interventions: Drug: DTG/ABC/3TC FDC DISPERSIBLE TABLET; Drug: EPZICOM (ABC/3TC); Drug: TIVICAY (DTG)
- SEQUENCE BCDEA (Experimental): Participants will receive treatment B in period 1, treatment C in period 2, treatment D in period 3, treatment E in period 4 and treatment A in period 5 (one treatment per period). Where A= EPZICOM (ABC 600 milligrams (mg)/3TC 300 mg) plus four TIVICAY (DTG 10 mg) tablets with ZMC water. B=Four TRIUMEQ (ABC 150mg/DTG 10 mg/3TC 75 mg) tablets dispersed in 40 mL stock solution 1 and consumed immediately. C=Four TRIUMEQ tablets dispersed in 40 mL stock solution 1, held for 30 mins, re-dispersed, and then consumed. D=Four TRIUMEQ tablets dispersed in 40 mL stock solution 2 and consumed immediately. E=Four TRIUMEQ tablets dispersed in 40 mL stock solution 2, held for 30 mins, re-dispersed, and then consumed.
  Interventions: Drug: DTG/ABC/3TC FDC DISPERSIBLE TABLET; Drug: EPZICOM (ABC/3TC); Drug: TIVICAY (DTG)
- SEQUENCE CDEAB (Experimental): Participants will receive treatment C in period 1, treatment D in period 2, treatment E in period 3, treatment A in period 4 and treatment B in period 5 (one treatment per period). Where A=EPZICOM (ABC 600 milligrams (mg)/3TC 300 mg) plus four TIVICAY (DTG 10 mg) tablets with ZMC water. B=Four TRIUMEQ (ABC 150mg/DTG 10 mg/3TC 75 mg) tablets dispersed in 40 mL stock solution 1 and consumed immediately. C=Four TRIUMEQ tablets dispersed in 40 mL stock solution 1, held for 30 mins, re-dispersed, and then consumed. D=Four TRIUMEQ tablets dispersed in 40 mL stock solution 2 and consumed immediately. E=Four TRIUMEQ tablets dispersed in 40 mL stock solution 2, held for 30 mins, re-dispersed, and then consumed.
  Interventions: Drug: DTG/ABC/3TC FDC DISPERSIBLE TABLET; Drug: EPZICOM (ABC/3TC); Drug: TIVICAY (DTG)
- SEQUENCE DEABC (Experimental): Participants will receive treatment D in period 1, treatment E in period 2, treatment A in period 3, treatment B in period 4 and treatment C in period 5 (one treatment per period). Where A=EPZICOM (ABC 600 milligrams (mg)/3TC 300 mg) plus four TIVICAY (DTG 10 mg) tablets with ZMC water. B=Four TRIUMEQ (ABC 150mg/DTG 10 mg/3TC 75 mg) tablets dispersed in 40 mL stock solution 1 and consumed immediately. C=Four TRIUMEQ tablets dispersed in 40 mL stock solution 1, held for 30 mins, re-dispersed, and then consumed. D=Four TRIUMEQ tablets dispersed in 40 mL stock solution 2 and consumed immediately. E=Four TRIUMEQ tablets dispersed in 40 mL stock solution 2, held for 30 mins, re-dispersed, and then consumed.
  Interventions: Drug: DTG/ABC/3TC FDC DISPERSIBLE TABLET; Drug: EPZICOM (ABC/3TC); Drug: TIVICAY (DTG)
- SEQUENCE EABCD (Experimental): Participants will receive treatment E in period 1, treatment A in period 2, treatment B in period 3, treatment C in period 4 and treatment D in period 5 (one treatment per period). Where A=EPZICOM (ABC 600 milligrams (mg)/3TC 300 mg) plus four TIVICAY (DTG 10 mg) tablets with ZMC water. B=Four TRIUMEQ (ABC 150mg/DTG 10 mg/3TC 75 mg) tablets dispersed in 40 mL stock solution 1 and consumed immediately. C=Four TRIUMEQ tablets dispersed in 40 mL stock solution 1, held for 30 mins, re-dispersed, and then consumed. D=Four TRIUMEQ tablets dispersed in 40 mL stock solution 2 and consumed immediately. E=Four TRIUMEQ tablets dispersed in 40 mL stock solution 2, held for 30 mins, re-dispersed, and then consumed.
  Interventions: Drug: DTG/ABC/3TC FDC DISPERSIBLE TABLET; Drug: EPZICOM (ABC/3TC); Drug: TIVICAY (DTG)

INTERVENTIONS:
Drug: DTG/ABC/3TC FDC DISPERSIBLE TABLET — DTG/ABC/3TC FDC dispersible tablet
Drug: EPZICOM (ABC/3TC) — EPZICOM will be available as orange, film coated, modified capsule shaped tablets, debossed with "GS FC2" on one side.
Drug: TIVICAY (DTG) — TIVICAY will be available as white, round, biconvex tablets

SUMMARY:
This is an open-label, randomized, crossover study in healthy adult subjects with 5 treatment groups over 5 dosing periods. This study will evaluate pharmacokinetic parameters and relative bioavailability of a dispersible, fixed-dose combination (FDC) tablet of TRIUMEQ™ ([abacavir, ABC]/[dolutegravir, DTG]/[lamivudine, 3TC]) when dispersed and consumed under four different dosing conditions in comparison to an oral dose of TIVICAY™ (DTG) + EPZICOM™ (ABC/3TC) non-dispersible tablets administered in the fasted state. Approximately 20 subjects will be randomized, each to one of 5 treatment groups. The total duration of participation of a subject in this study will be approximately 10-11 weeks. It will include a screening visit within 30 days prior to the first dose of study drug, five treatment periods each with a single dose of study drug per treatment period and a follow up visit within 7 10 days after the last dose. There will also be a washout of at least 7 days between doses in each treatment period. TRIUMEQ, EPZICOM, and TIVICAY are trademarks of the GlaxoSmithKline group of companies.

ELIGIBILITY:
Inclusion Criteria

* Male or female aged between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac evaluation (history and ECG). A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilogram (kg) for males and >=45 kg for females and body mass index (BMI) within the range 18.5-31.0 kg/m^2 (inclusive).
* Male or female
* Females of non-reproductive potential defined as pre-menopausal females with documented tubal ligation, documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion, hysterectomy, documented bilateral oophorectomy, postmenopausal defined as 12 months of spontaneous amenorrhea (in questionable cases a blood sample with simultaneous follicle stimulating hormone [FSH] and estradiol levels consistent with menopause). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.
* Female of reproductive potential and agrees to follow one of the options listed in the Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) from 30 days prior to the first dose of study medication and until 2 weeks after dosing with study medication and completion of the follow-up visit. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.
* Documentation that the subject is negative for the human leukocyte antigen (HLA)-B*5701 allele.

Exclusion Criteria

* ALT and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) >450 milliseconds (msec). The specific formula that will be used to determine eligibility and discontinuation for an individual subject should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual subject and then the lowest QTc value used to include or discontinue the subject from the trial.
* Unable to refrain from the use of prescription (i.e., dofetilide) or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 gram of alcohol: 12 ounces (360 mL) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 1 month prior to screening.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Creatinine clearance (CrCL) <60 mL/min
* Presence of HBsAg, positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* Where participation in the study would result in donation of blood or blood product in excess of 500 mL within 56 days.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-09-01; Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-25 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUC[0-infinity]) of DTG, ABC, and 3TC | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48 and 72 h post dose
  Blood samples will be collected at pre-dose and at specific post-dose time points for calculating AUC [0- infinity]
Maximum observed plasma concentration (Cmax) of DTG, ABC, and 3TC | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48 and 72 h post dose
  Blood samples will be collected at pre-dose and at specific post dose time points for calculating Cmax

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve from time zero (pre-dose) to 24 hours (h) AUC(0-24) of DTG, ABC, and 3TC | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24h post dose in each of the 5 treatment periods.
  AUC(0-24) is defined as the area under the concentration-time curve from time zero (pre-dose) to 24 h post-dose.
Area under the plasma concentration-time curve from time zero (pre-dose) to time of last measurable concentration (AUC[0 t]) of DTG, ABC, and 3TC | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48 and 72 h post dose in each of the 5 treatment periods.
  Blood samples will be collected at pre-dose and at specific post dose time points for calculating AUC [0-t]
Time to maximum plasma concentration (Tmax) of DTG, ABC, and 3TC | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48 and 72 h post dose in each of the 5 treatment periods.
  Blood samples will be collected at pre-dose and at specific post-dose time points for calculating Tmax
Apparent clearance following oral dosing (CL/F) of DTG, ABC, and 3TC | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48 and 72 h post dose in each of the 5 treatment periods.
  Blood samples will be collected at pre-dose and at specific post-dose time points for calculating CL/F
Concentration at 24 h after dose administration (C24) of DTG, ABC, and 3TC | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24h post dose in each of the 5 treatment periods.
  Blood samples will be collected at pre-dose and at specific post-dose time points for calculating C24
Terminal phase half-time (t1/2) of DTG, ABC, and 3TC | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48 and 72 h post dose in each of the 5 treatment periods.
  Blood samples will be collected at pre-dose and at specific post-dose time points for calculating t1/2
Absorption lag time (Tlag) of DTG | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 48 and 72 h post dose in each of the 5 treatment periods.
  Absorption lag time is defined as the time taken for a drug to appear in the systemic circulation following administration
Number of subjects with adverse event (AE) and serious adverse event (SAE). | Approximately 11 weeks
  AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment will be categorized as SAE.
Blood pressure assessment as a safety measure | Approximately 11 weeks
  Systolic and diastolic blood pressure will be measured in supine or semi-supine position after 5 minutes rest at Day -1, pre-dose, 4h, 24h, 48 h, 72h post-dose, and at follow up
Measurement of pulse rate as a safety measure | Approximately 11 weeks
  Heart rate will be measured at supine or semi-supine position after 5 minutes rest at Day -1, pre-dose, 4h, 24h, 48 h, 72h post-dose, and at follow up
Body temperature assessment as a safety measure | Approximately 11 weeks
  Temperature will be recorded at supine or semi-supine position after 5 minutes rest at Day -1, pre-dose, 4h, 24h, 48 h, 72h post-dose, and at follow up
Electrocardiogram (ECG) assessment as a measure of safety | Approximately 11 weeks
  Single 12-lead ECGs will be obtained in a supine or semi-supine position having rested in this position for at least 10 minutes beforehand at Day -1 of each of 5 treatment periods
Number of subjects having abnormal clinical laboratory parameters as a measure of safety | Approximately 11 weeks
  Blood samples will be collected (at Day -1, and 24 h post-dose and at follow-up if needed) to analyze blood urea nitrogen, creatinine, glucose, creatine phosphokinase (CPK), sodium, potassium, calcium, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), total bilirubin, direct bilirubin, total protein, albumin
Number of subjects having abnormal hematology laboratory parameters as a measure of safety | Approximately 11 weeks
  Blood samples will be collected (at Day -1 and 24h post-dose and at follow-up if needed) to analyze platelet count, Red Blood Cells (RBC) count, hemoglobin, hematocrit, mean corpuscular volume ( MCV), mean corpuscular hemoglobin (MCH) White Blood Cells (WBC), neutrophils, lymphocytes, monocytes, eosinophils, and basophils
Number of subjects having abnormal urinalysis as a measure of safety | Approximately 11 weeks
  Urine samples will be collected (at Day -1, and 24 h post-dose and at follow-up if needed) to analyze specific gravity, pH, glucose, protein, blood and ketones by dipstick, and for microscopic examination

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Singh RP, Shaik JSB, Skoura N, Joshi S, Shreeves T, Casillas L, Buchanan AM. Effects of Low- and High-Mineral Content Water on the Relative Bioavailability of a Coformulated Abacavir/Dolutegravir/Lamivudine Dispersible Tablet in Healthy Adults. J Acquir Immune Defic Syndr. 2018 Dec 15;79(5):631-638. doi: 10.1097/QAI.0000000000001859. PMID 30239425